CLINICAL TRIAL: NCT06808529
Title: A Study on the Effectiveness of Pilates and TENS Acupuncture in Treating Primary Dysmenorrhea in Female Students At King Aboulaziz University (KAU)
Brief Title: Effect of Pilates Exercises and TENS Acupuncture in Primary Dysmenorrhea Among Female Students At KAU
Acronym: KAU
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Mohamed Elnahas, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMRS-EC2024-030
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Dysmenorrhea Primary
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Pilates exercises and TENS Acupuncture
  Interventions: Device: Pilates exercises and TENS Acupuncture
- Control group (Experimental): Conservative treatment
  Interventions: Drug: ibuprofen 400 mg

INTERVENTIONS:
Device: Pilates exercises and TENS Acupuncture — All performed Pilates exercises for 24 session, 3 sessions per week for (2 consecutive menstrual cycle), each session lasted for 30 minutes in addition to application of TENS acupuncture therapy for 30 minutes, 3 sessions in the first 3 days for (2 consecutive menstrual cycle).
  Arms: Study group
Drug: ibuprofen 400 mg — All took capsules of ibuprofen(400-milligram) and instructed to take them once every eight hours for three days, one day before the start of their menstrual cycle and on the first two days of menstruation for (2 consecutive menstrual cycle).
  Arms: Control group

SUMMARY:
This study was done to determine the effect of Pilates exercises and TENS acupuncture in primary dysmenorrhea among female students at King Abdulaziz University (KAU).

ELIGIBILITY:
Inclusion Criteria:

* Participants suffering from primary dysmenorrhea.
* Their age ranged between 18-24 years
* Their BMI less than 30 kg/m2.

Exclusion Criteria:

* Gynecological disorders (secondary dysmenorrhea)
* Married females,
* Low back pain due to any other pathology
* Chronic diseases (diabetes, high blood pressure)

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Primary dysmenorrhea.
Enrollment: 30 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue scale | 2 months
  Visual Analogue scale for assessing pain level, a score ranging from 0 to 100 mm.

SECONDARY OUTCOMES:
Verbal multidimensional scoring system of dysmenorrhea | 2 months
  * Grade 0: The menstrual cycle causes no pain and has no effect on day-to-day activities.
  * Grade 1: Although uncomfortable menstruation never gets in the way of a woman's regular activities, and analgesics are rarely needed.
  * Grade 2 : daily activities are disrupted and analgesics have a poor effect .
  * Grade 3: Activity is obviously impeded, analgesics have a poor effect and symptoms such as headache, fatigue, nausea, vomiting, and diarrhea is present

CONTACTS AND LOCATIONS:
Locations (1):
- king Abdulaziz university, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: article — https://pubmed.ncbi.nlm.nih.gov/21799683/